CLINICAL TRIAL: NCT03894683
Title: Effect of Melatonin on Cardiovascular and Muscle Function in Patients With Heart Failure: a Double Blinded Prospective Randomized Clinical Trial.
Brief Title: Effect of Melatonin on Cardiovascular and Muscle Mass and Function in Patients With Heart Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Collaborators: National Institute for Medical Research Development (Unknown)
Responsible Party: Principal Investigator, Masoumeh Sadeghi, Head of Cardiac Rehabilitation Research Center, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 397180
Record Dates: First submitted 2019-03-27; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Heart failure; Melatonin; Muscle wasting
MeSH Terms: conditions — Heart Failure; Muscular Atrophy | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin (Experimental): Melatonin (10 mg tablets) by oral root, ingested at bedtime for 6 months
  Interventions: Drug: Melatonin 10 mg
- Placebo (Placebo Comparator): Placebo tablets in the same shape as melatonin tablets, ingested the same as the melatonin tablets.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Melatonin 10 mg — Melatonin tablets (10 mg)
  Arms: Melatonin
Drug: Placebo Oral Tablet — Placebo tablets manufactured the same as melatonin tablets
  Arms: Placebo

SUMMARY:
The main aim of this study is to investigate the effect of melatonin on clinical outcome, quality of life, and cardiovascular function of the patients with heart failure, as well as its effect on their skeletal muscle mass and function.

DETAILED DESCRIPTION:
People with heart failure (HF) suffer from various comorbidities and complications which their management is as important as treatment of HF per se. An important complication of the HF is progressive decrease in muscle mass and function known as muscle wasting or sarcopenia. Prevention, diagnosis, and treatment of muscle wasting is emphasized to improve prognosis and quality of life of the patients with HF. Melatonin is a natural hormone which is secreted from pineal gland and is involved in circadian rhythm control. Recent data delineates more important roles for melatonin in cellular metabolism and apoptosis, as well as acting as an antioxidant and anti-inflammatory agent in the body. Experimental studies show that melatonin can have a beneficial role in muscle wasting in several chronic conditions such as heart failure. Furthermore melatonin has been shown to have valuable effects on cardiovascular health, blood pressure, and endothelial function and it might benefit patients with heart failure. In this study the effect of melatonin on clinical outcome and quality of life of the patients with HF and their echocardiographic parameters, muscle mass, muscle function, inflammatory biomarkers, serum metabolic parameters, and serum oxidative stress markers will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Systolic heart failure with ejection fraction < 40, either ischemic or dilated cardiomyopathy (DCM)
* Symptoms and medications of HF have been stable for at least three months
* NYHA class II-III
* Willing to participate in the study and providing informed consent

Exclusion Criteria:

* Chronic comorbidities: insulin dependent diabetes, renal failure (GFR < 30 mL/min per 1.73 m2), uncontrolled endocrine disease, end-stage liver disease, rheumatological disease, chronic obstructive pulmonary disease (class D according to GOLD classification), morbid obesity (BMI > 35)
* Acute ischemic heart event or revascularization procedure in the last month
* Regular supervised exercise or ingestion of muscle hypertrophy supplementations in the last three months
* Vegetarian diet or sever restriction of protein in the diet in the last three months
* Occurrence of melatonin related adverse effects

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Composite clinical endpoint score | 6 months or earlier if patient was dropped out from the study
  A score with the following components: all-cause mortality, hospitalization for heart failure during the study, and change in quality of life by Minnesota Living with Heart Failure Questionnaire (MLHFQ)

SECONDARY OUTCOMES:
Adverse effects of melatonin | Throughout the study up to 6 months
  Adverse effects detected in the melatonin group compared with the placebo group
Change in appendicular lean mass (kg) | Baseline and 6 months
  Measured by dual-energy x-ray absorptiometry
Change in lean body mass (kg) | Baseline and 3 months
  Measured by bioimpedance analysis
Change in lean body mass (kg) | Baseline and 6 months
  Measured by bioimpedance analysis
Change in grip strength (kg) | Baseline and 3 months
  Measured by a hydraulic dynamometer
Change in grip strength (kg) | Baseline and 6 months
  Measured by a hydraulic dynamometer
Change in exercise capacity | Baseline and 3 months
  Measured by 6 minute walk test
Change in exercise capacity | Baseline and 6 months
  Measured by 6 minute walk test
Change in Left ventricular ejection fraction (LVEF) | Baseline and 6 months
  Measured by echocardiography using the Simpson method
Change in left ventricular end-systolic volume (LVESV) | Baseline and 6 months
  Measured by echocardiography using the Simpson method
Change in endothelial dysfunction | Baseline and 6 months
  Measured by flow-mediated vasodilation (FMD) method
Change in mean systolic and diastolic blood pressures | Baseline and 3 months
  Mean of two measurements, using an automated electronic oscillometric device
Change in mean systolic and diastolic blood pressures | Baseline and 6 months
  Mean of two measurements, using an automated electronic oscillometric device

OTHER OUTCOMES:
Change in fasting blood glucose level (mg/dl) | Baseline and 6 months
  Measured in serum samples after 12h fasting
Change in serum lipid levels (mg/dl) | Baseline and 6 months
  Including triglyceride, LDL, and HDL, measured in serum samples after 12h fasting
Change in serum insulin, and IGF-1 levels | Baseline and 6 months
  Measured by enzyme-linked immunosorbent assay (ELISA) on serum samples stored at -80°
Change in level of serum inflammatory biomarkers | Baseline and 6 months
  Measured by enzyme-linked immunosorbent assay (ELISA) on serum samples stored at -80°
Change in level of serum oxidative stress biomarkers | Baseline and 6 months
  Including malondialdehyde (MDA) and total antioxidant capacity (TAC)
Changes in psychological status of the patients | Baseline and 6 months
  Including anxiety (by Spielberger State - Trait Anxiety Inventory (STAI)) and depression (by Beck Depression Inventory)
Changes in sleep quality of the patients | Baseline and 6 months
  Measured by Pittsburgh Sleep Quality Index (PSQI) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Masoumeh Sadeghi, MD, Principal Investigator — Cardiac Rehabilitation Research Center
Locations (1):
- Cardiac rehabilitation research center, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Six months after publication